CLINICAL TRIAL: NCT00004640
Title: Trials to Enhance Elders' Teeth and Oral Health
Brief Title: "Clinical Trials to Enhance Elders' Oral Health" ("TEETH")
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIDCR-008; R01DE012215 (NIH)
Record Dates: First submitted 1999-09-17; First posted 1999-09-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Tooth Loss; Periodontal Disease; Tooth Decay
Keywords: Aging; Elderly; Periodontal Disease; Dental Caries; Fluoride; Antibacterial rinse; Chlorhexidine; Tooth Mortality
MeSH Terms: conditions — Tooth Loss; Periodontal Diseases; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Chlorhexidine rinse — chlorhexidine solution on tooth loss in low income

SUMMARY:
The purpose of this study is to determine if regular rinsing with chlorhexidine is effective as a long-term preventive method for reducing the incidence of tooth loss in low income older adults. The true end-point of the study is tooth loss after five years of regular rinsing with chlorhexidine or a placebo; surrogate endpoints are periodontal disease, root and coronal decay.

DETAILED DESCRIPTION:
"TEETH" is a double-blinded, randomized clinical trial, supervised by a Data & Safety Monitoring Board, designed to provide unequivocal evidence regarding the impact of regular rinsing 0.12% chlorhexidine solution on tooth loss in low income, community-dwelling older adults who are irregular users of dental services. Of the 1101 subjects enrolled in the study in Seattle, WA and Vancouver, B.C., one/half have been assigned to the active rinse condition; the other half to the placebo rinse which looks and tastes like the chlorhexidine rinse but does not have the active ingredient. Subjects receive two bottles of rinse every six months; the first to be used daily for one month, the second weekly for five months. Reminder calls are designed to help subjects maintain this rinse regimen. Subjects return yearly to research clinics at each participating university, where they are examined by a dentist who is trained in clinical research methodology and calibrated annually. The purpose of these visits is to examine subjects for tooth loss (followed by contacts with extracting dentists to determine the dentist's reasons for extracting the tooth), pocket depth, recession, caries and restorations on root and coronal surfaces. Interviews are also conducted annually with participants to assess health status, health behaviors, and oral health quality of life. A panoramic radiograph was taken at baseline of each subject and is to be done again at the five-year (final) yearly exam. These radiographs are used to confirm tooth loss and possible reasons for extractions

ELIGIBILITY:
Inclusion Criteria:

* Age at entry 60-75
* Four or more natural teeth
* No preventive dental visits in the past 18 months
* Scores > or = 60 on a measure of oral health self-efficacy (max possible=100)
* willing to participate in a five-year study
* willing to use rinses on a prescribed regimen and to return for yearly cleaning and exam appointments.

Exclusion criteria:

* Not having a phone at home for follow-up calls

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1101 (Estimated)
Dates: Start 1998-05; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
regular rinsing with chlorhexidine is effective method for reducing the incidence of tooth loss in low income older adults. | five years of regular rinsing

CONTACTS AND LOCATIONS:
Locations (2):
- University of Washington, Seattle, Washington, United States
- University of British Columbia, Vancouver, British Columbia, Canada